CLINICAL TRIAL: NCT06817018
Title: Ginger and the Microbiota-gut-brain Connection in Sciatic Pain Individuals
Brief Title: Ginger Root Extract for Sciatic Pain Individuals
Acronym: Ginger-NP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Leslie Shen (Other)
Responsible Party: Sponsor-Investigator, Leslie Shen, Professor of Pathology, Texas Tech University Health Sciences Center
Organization: Texas Tech University Health Sciences Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ginger-sciatic pain
Record Dates: First submitted 2025-02-03; First posted 2025-02-10 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Neuropathic Pain; Sciatic Pain
MeSH Terms: conditions — Neuralgia | interventions — ginger extract

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo group: 2,000 mg cellulose daily for 8 weeks
  Interventions: Dietary Supplement: Placebo
- Ginger (Active Comparator): Ginger group: 2,000 mg ginger root extract daily for 8 weeks
  Interventions: Drug: Ginger

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo (Sabinsa)
  Arms: Placebo
Drug: Ginger — Ginger root extract
  Arms: Ginger

SUMMARY:
Neuropathic pain affects the quality of life of many Americans. Non-pharmacological strategies such as bioactive compounds in foods are being explored as therapeutics but can also serve as tools to better understand pain mechanisms. The previous study reported that ginger root extract supplementation palliated pain-spectrum behaviors in animals with neuropathic pain via the microbiota-gut-brain axis. The proposed study is primarily designed to use ginger supplementation for a better understanding of the role of microbiota-gut-brain interactions in sciatica states in a randomized, double-blinded, and placebo-controlled trial. Eighty participants with sciatica will be randomized to receive placebo (2000 mg starch daily) or ginger (2000 mg daily) for 8 weeks. This study will evaluate the effects of ginger supplementation on gut function measured as gut microbiota composition using 16S rRNA sequencing analysis, intestinal permeability based on plasma lipopolysaccharide binding protein and fecal zonulin using ELISA, and fecal metabolites using LC-MS/MS analysis (SA 1); on neuroinflammation in whole blood mRNA using nCounter® Neuroinflammation Panels analysis (SA 2); and on pain-associated outcomes and brain neuroplasticity by assessing functional (resting state-fMRI) and structural (Diffusion Tensor Imaging) connectivity (SA 3).

ELIGIBILITY:
Inclusion criteria:

* 18-85 years old men and women with BMI < 25 or ≥ 30 kg/m2
* low back or gluteal pain radiating into leg(s) past the knee (sciatica) with pain duration of at least 3 months (chronic sciatica)
* pain scale > 3 out of 10 (0=no pain,10=worst pain imaginable) during the past 24 hours
* willingness to accept randomization.
* woman of childbearing potential agrees to use an effective form of contraception during the study

Exclusion criteria:

Sciatica aspects:

* known or suspected serious spinal pathology (e.g., cauda equina syndrome or spinal fracture)
* scheduled, or being considered, for spinal surgery or interventional procedures for sciatica during study period
* focal neurological deficits with progressive or disabling symptoms
* low back pain without sciatica

GI aspects:

* unstable GI disorder
* history of chronic or systemic autoimmune diseases with GI involvement
* recent (<1 month) appearance of diarrhea or hematochezia before study begins
* recent (<1 month) exposure to antibiotics before study start

Other exclusion considerations:

* pregnant or breast-feeding women
* women of child-bearing potential will have a urine pregnancy test done prior to the baseline MRI and administration of any study drug. The clinical research coordinator will run the pregnancy test and inform the patient of the results. If the test is positive, they will be withdrawn from study participation.
* cognitive impairment, history of psychiatric conditions indicating mental health instability or incapacity
* likeliness of moving during the trial, lack of transportation, or unavailability at sample collection times.
* presence of a bleeding diathesis
* taking anticoagulant medications (e.g Heparin, Warfarin)
* taking dual antiplatelet medications (e.g. aspirin + Plavix)
* participants with clinically significant laboratory abnormalities of liver function (AST and ALT) and kidney function (BUN and serum creatinine) abnormalities. Definition of clinically significant for liver function is AST/ALT ≥ 3.0x ULN and for kidney function is serum creatinine > 2.0 mg/dl and BUN > 1.5x ULN.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
plasma lipopolysaccharide binding protein (LBP) | baseline and after 8 weeks
  Intestinal permeability biomarker
fecal zonulin | baseline and after 8 weeks
  intestinal permeability marker
brief pain inventory (BPI) | baseline and after 8 weeks
  pain assessment
SF-MPQ | baseline and after 8 weeks
  pain assessment

SECONDARY OUTCOMES:
fecal metabolites using LC-MS/MS analysis | baseline and after 8 weeks
  Untargeted fecal metabolites will be assessed using LC-MS/MS analysis and the combination of retention time and mass signature provides great specificity for each metabolite identification.
gut microbiome using 16S rRNA amplicon sequencing | baseline and after 8 weeks
  Fecal gut microbiome composition is a collection of microorganisms that live in the human digestive tract.
neuroinflammation genes | baseline and after 8 weeks
  Whole blood neuroinflammation gene profiles will be analyzed using nCounter® Neuroinflammation Panel to evaluate pathways, processes, and cell types that are involved in neuroinflammation.
structural connectivity using resting state-fMRI | baseline and after 8 weeks
  Resting state-fMRI connectivity in brain will be examined between the left and right amygdala seed regions and the broader bilateral mPFC, defined using the probabilistic Harvard-Oxford Subcortical Structural Atlas in FSL.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available due to HIPAA regulation.

REFERENCES:
- [Background] Shen CL, Watkins BA, Kahathuduwa C, Chyu MC, Zabet-Moghaddam M, Elmassry MM, Luk HY, Brismee JM, Knox A, Lee J, Zumwalt M, Wang R, Wager TD, Neugebauer V. Tai Chi Improves Brain Functional Connectivity and Plasma Lysophosphatidylcholines in Postmenopausal Women With Knee Osteoarthritis: An Exploratory Pilot Study. Front Med (Lausanne). 2022 Jan 3;8:775344. doi: 10.3389/fmed.2021.775344. eCollection 2021. PMID 35047525
- [Background] Goncalves L, Dickenson AH. Asymmetric time-dependent activation of right central amygdala neurones in rats with peripheral neuropathy and pregabalin modulation. Eur J Neurosci. 2012 Nov;36(9):3204-13. doi: 10.1111/j.1460-9568.2012.08235.x. Epub 2012 Aug 3. PMID 22861166
- [Background] Checchia GA, Letizia Mauro G, Morico G, Oriente A, Lisi C, Polimeni V, Lucia M, Ranieri M; Management of Peripheral Neuropathies Study Group. Observational multicentric study on chronic sciatic pain: clinical data from 44 Italian centers. Eur Rev Med Pharmacol Sci. 2017 Apr;21(7):1653-1664. PMID 28429339
- [Background] Nation KM, De Felice M, Hernandez PI, Dodick DW, Neugebauer V, Navratilova E, Porreca F. Lateralized kappa opioid receptor signaling from the amygdala central nucleus promotes stress-induced functional pain. Pain. 2018 May;159(5):919-928. doi: 10.1097/j.pain.0000000000001167. PMID 29369967
- [Background] U Jumbo S, C MacDermid J, E Kalu M, L Packham T, S Athwal G, J Faber K. Measurement Properties of the Brief Pain Inventory-Short Form (BPI-SF) and the Revised Short McGill Pain Questionnaire-Version-2 (SF-MPQ-2) in Pain-related Musculoskeletal Conditions: A Systematic Review Protocol. Arch Bone Jt Surg. 2020 Mar;8(2):131-141. doi: 10.22038/abjs.2020.36779.1973. PMID 32490042
- [Background] Dworkin RH, Turk DC, Revicki DA, Harding G, Coyne KS, Peirce-Sandner S, Bhagwat D, Everton D, Burke LB, Cowan P, Farrar JT, Hertz S, Max MB, Rappaport BA, Melzack R. Development and initial validation of an expanded and revised version of the Short-form McGill Pain Questionnaire (SF-MPQ-2). Pain. 2009 Jul;144(1-2):35-42. doi: 10.1016/j.pain.2009.02.007. Epub 2009 Apr 7. PMID 19356853
- [Background] Shen CL, Wang R, Ji G, Elmassry MM, Zabet-Moghaddam M, Vellers H, Hamood AN, Gong X, Mirzaei P, Sang S, Neugebauer V. Dietary supplementation of gingerols- and shogaols-enriched ginger root extract attenuate pain-associated behaviors while modulating gut microbiota and metabolites in rats with spinal nerve ligation. J Nutr Biochem. 2022 Feb;100:108904. doi: 10.1016/j.jnutbio.2021.108904. Epub 2021 Nov 6. PMID 34748918
- [Background] Shen CL, Wang R, Yakhnitsa V, Santos JM, Watson C, Kiritoshi T, Ji G, Hamood AN, Neugebauer V. Gingerol-Enriched Ginger Supplementation Mitigates Neuropathic Pain via Mitigating Intestinal Permeability and Neuroinflammation: Gut-Brain Connection. Front Pharmacol. 2022 Jul 8;13:912609. doi: 10.3389/fphar.2022.912609. eCollection 2022. PMID 35873544